CLINICAL TRIAL: NCT05796050
Title: Sex Related Differences in Systolic and Diastolic Cardiac Function in Dependence From Lifestyle Modification Factors
Brief Title: Sex Related Differences in Cardiac Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-1812
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Diastolic Dysfunction; Systolic Dysfunction
Keywords: Sex-Related differences cardiovascular disease; Cardiovascular Disease; Transthoracic echocardiography; myocardial strain; cardiomyopathies
MeSH Terms: conditions — Cardiovascular Diseases; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to investigate sex-specific differences in LV and RV function (systolic and diastolic) with regarding the development and progression of heart failure with preserved ejection fraction based on a retrospective data analysis. Lifestyle modification factors will be assessed for multivariate analyses in order to detect influencing factors. Progression will be analysed in a retrospective time series analysis.

DETAILED DESCRIPTION:
Compared to men, women show a different cardiovascular risk profile, In this context, it has already been shown that mortality in women with cardiovascular diseases is increased. Along with this, there are first indications of an echocardiographic altered cardiac function. It was shown that women are more prone to heart failure with preserved ejection fraction. However, the underlying mechanisms and driving factors have not yet been fully explored. Moreover, the role of associated factors such as smoking, bodyweight or cardiovascular risk factors and menopause status remain nut fully understood.

In this project differences differences in sex-specific LV and RV function depending on defined risk factors will be investigated. For this purpose, a retrospective follow-up analysis willl be carried out. This is based on test results from patients who underwent transthoracic echocardiography in the echocardiography department of the Department of Cardiology, Pneumology and Angiology University Hospital Düsseldorf.

The aim is to evaluate possible differences in the sex-specific risk profile. This may allow us to define the cardiovascular risk profile in dependence from each sex more concretely.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent at least one transthoracic echocardiography in between 2019-2022

Exclusion Criteria:

* < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that underwent transthoracic echocardiography in the department of Cardiology, Pneumology and Vascular Medicine, University Hospital Düsseldorf.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2022-02-02 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Occurence of Heart Failure with preserved ejection fraction | 3 years
  measured by transthoracic echocardiography

SECONDARY OUTCOMES:
Change in ejection fraction | 3 years
  measured by transthoracic echocardiography
Changes in Myocardial strain analysis | 3 years
  measured by transthoracic echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Malte Kelm, Prof., Study Chair — Clinic for Cardiology, Pneumology and Angiology at University Hospital Düsseldorf
Locations (1):
- University-Hospital Düsseldorf Division of Cardiology, Pulmonary Disease and Vascular Medicine, Düsseldorf, Germany